CLINICAL TRIAL: NCT02938962
Title: Revision Total Hip Arthroplasty: Comparison of the Effects of Intravenous and Topically Administered Tranexamic Acid in a Prospective Randomized Trial (VITALITY-X)
Brief Title: Intravenous vs. Topical Tranexamic Acid in Revision THA (VITALITY-X)
Acronym: VITALITY-X
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mount Sinai Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 16-0046-A
Record Dates: First submitted 2016-10-03; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Tranexamic Acid; Blood Loss, Surgical; Arthroplasty, Replacement, Hip
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intravenous TXA (Active Comparator): The IV administration group will receive a single 20mg/kg dose of TXA prior to the skin incision.
  Interventions: Drug: Tranexamic Acid
- Topical TXA (Active Comparator): The topical administration group will have a 100mL solution (3g TXA in 100cc of normal saline) instilled into the surgical field throughout the operative procedure; 50mL of the solution will be instilled after bony preparation of the acetabulum and/or femur and 50mL of the solution will be instilled prior to closure. The topical TXA solution will be allowed to bathe the wound for 5 minutes at each administration.
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid

SUMMARY:
The objective of this study is to evaluate and compare the effects of intravenous and topical administration of tranexamic acid during revision hip arthroplasty on blood loss, allogenic blood transfusion rates, length of hospital stay and perioperative complications.

DETAILED DESCRIPTION:
This study will use a prospective randomized single-blinded study design. The study will include one hundred and sixty patients undergoing revision total hip arthroplasty at a single institution (Mount Sinai Hospital (MSH), Toronto, ON, Canada). Tranexamic acid has been routinely administered as a single intravenous preoperative dose (unless contraindicated) in all revision hip arthroplasty cases at MSH since May 2012. In this study, participants will be randomized into 2 treatment groups: intravenous (IV) administration of tranexamic acid (TXA) and topical administration of TXA. The IV administration group will receive a single 20mg/kg dose of TXA prior to the skin incision. The topical administration group will have a 100mL solution (3g TXA in 100cc of normal saline) instilled into the surgical field during surgery. The primary outcome measured will be the delta hemoglobin (defined as the change in hemoglobin from preoperative measurement to POD 0, 1, 2, 3, 5). Secondary outcomes to be analyzed include intraoperative estimated blood loss, allogenic blood transfusion rates, length of hospital stay and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of surgery.
* Consent for transfusion of blood or blood-related products.
* No contraindication to use of tranexamic acid.
* Revision hip arthroplasty performed at MSH.
* Indication for surgery including osteolysis, component failure, prosthetic joint infection, aseptic/septic loosening, periprosthetic fracture, recurrent instability/dislocation, polyethylene wear and abductor insufficiency.
* Revision hip arthroplasty procedure performed including acetabular component revision, femoral component revision, impaction bone grafting, proximal femoral allograft, proximal femoral replacement, removal of hardware (excluding head/liner exchanges).
* Direct lateral (transgluteal, Hardinge) approach utilized, including augmentation with extended trochanteric osteotomy (ETO), trochanteric slide and modified trochanteric slide.

Exclusion Criteria:

* Age < 18 years at the time of surgery.
* Posterior (Moore, Southern) or Anterior (Smith-Peterson) operative approach utilized.
* Implantation of surgical drain.
* Patients undergoing any isolated combination of femoral head exchange, acetabular liner exchange and abductor repair.
* Patients with an absolute contraindication to tranexamic acid use including:
* Allergy to TXA or previous adverse reaction to TXA/its constituents.
* Thrombolytic events <1 year prior to surgery (myocardial infarction, cerebrovascular accident, pulmonary embolus).
* Active thrombolytic event and/or on lifelong anticoagulant.
* Known coronary artery disease.
* Renal failure with serum creatinine >200µmol/L, creatinine clearance <50mL/min and/or dialysis patient.
* Patients with disseminated intravascular coagulation.
* Patients currently using Oral Contraceptive medication.
* Patients with a relative contraindication to tranexamic acid use deemed inappropriate for tranexamic acid administration by Anesthesiology team, including:
* Thrombolytic events >1 year prior to surgery (myocardial infarction, cerebrovascular accident, pulmonary embolus).
* History of cancer.
* Patients with a history of acquired disturbances in color vision.
* Clinical judgment by Anesthesiology team not otherwise specified.
* Patients ineligible or refusing to consent for allogenic blood transfusion.
* Blood conservation augmentation strategies utilized:
* Cell saver/autotransfusion.
* Administration of erythropoietin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Delta Hemoglobin | Post-operative day #0 to post-operative day #5
  Delta hemoglobin (defined as the change in hemoglobin from preoperative measurement to post-operative day 0, 1, 2, 3, 5).

SECONDARY OUTCOMES:
Allogenic blood units transfused | through hospital admission, an average of 4 days
Length of stay | through hospital admission, an average of 4 days
Estimated intra-operative blood loss as assessed by the anaesthesiology team | Intra-operative
Post-operative complications | 3 months postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kuzyk, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada